CLINICAL TRIAL: NCT01673035
Title: Cognitive Behavior Therapy vs. Behavioral Stress Management for Severe Health Anxiety: a Randomized Controlled Trial of Two Internet-based Treatments
Brief Title: Internet Treatment for Health Anxiety
Acronym: HA-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA-X
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Hypochondriasis
MeSH Terms: conditions — Hypochondriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- internet-based CBT (Experimental): Cognitive behavior therapy delivered via the internet: 12 weeks, therapist-guided
  Interventions: Behavioral: CBT, exposure and response prevention
- internet-based BSM (Active Comparator): behavioral stress management delivered via the internet: 12 weeks, therapist-guided
  Interventions: Behavioral: BSM, stress management and applied relaxation

INTERVENTIONS:
Behavioral: CBT, exposure and response prevention — This intervention entails different exercises aimed exposure to health anxiety stimuli.
  Arms: internet-based CBT
Behavioral: BSM, stress management and applied relaxation — BSM, this intervention comprises structured exercises aimed at reducing stress and controlling the anxiety response. One main component is applied relaxation.
  Arms: internet-based BSM

SUMMARY:
Background

Severe health anxiety, hypochondriasis according to DSM-IV, is common and associated with functional disability. Cognitive behavior therapy (CBT) and behavioral stress management (BSM) have been showed to be effective in the treatment of severe health anxiety. The mechanisms of the treatments are however poorly understood. In addition, effective psychological treatments are accessible to only a few. One prior RCT has shown that internet-based CBT could be effective in comparison to waiting list controls. More studies on internet-based CBT is essential to establish evidence. In addition, few studies with sufficient power have investigated the effect of CBT in comparison to other active treatments.

Aim of the study The aim of the present RCT is to compare internet-based CBT (n=110) to behavioral stress management (n=110) for adult participants with severe health anxiety. BSM is considered a comparison treatment for two reasons: it has been shown to be effective and it lacks exposure and response prevention, which is suggested to be an important mechanism in CBT.

Participants in both treatments are expected to be significantly improved on measures of health anxiety. Participants receiving CBT are expected to be significantly more improved compared to participants receiving BSM.

DETAILED DESCRIPTION:
Background

Severe health anxiety, hypochondriasis according to DSM-IV, is common and associated with functional disability. Cognitive behavior therapy (CBT) and behavioral stress management (BSM) have been showed to be effective in the treatment of severe health anxiety. The mechanisms of the treatments are however poorly understood. In addition, effective psychological treatments are accessible to only a few. One prior RCT has shown that internet-based CBT could be effective in comparison to waiting list controls. More studies on internet-based CBT is essential to establish evidence. In addition, few studies with sufficient power have investigated the effect of CBT in comparison to other active treatments.

Aim of the study The aim of the present RCT is to compare internet-based CBT (n=110) to behavioral stress management (n=110) for adult participants with severe health anxiety. BSM is considered a comparison treatment for two reasons: it has been shown to be effective and it lacks exposure and response prevention, which is suggested to be an important mechanism in CBT.

The investigators expect participants in both treatments to be significantly improved on measures of health anxiety. Participants receiving CBT are expected to be significantly more improved compared to participants receiving BSM.

Design:

Randomized controlled trial. Participants are randomized in a 1:1 ratio.

Assessments:

The primary outcome measure is the Health Anxiety Inventory (HAI). Assessments with HAI are conducted at baseline, post-treatment, 3- and 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of severe health anxiety (hypochondriasis) according to DSM-IV
* At least 18 years old
* Able to read and write in Swedish

Exclusion Criteria:

* Other primary axis-I disorder
* Ongoing substance abuse or addiction
* current or previous episode of psychosis or bipolar disorder
* higher score than 30 on the Montgomery åsberg depression rating scale-self report
* higher than 3 on the suicide item of the MADRS-S
* non-stable antidepressant medication during last 2 months if on this kind of medication
* ongoing concurrent psychological treatment for severe health anxiety
* having received previous high quality CBT during the recent 3 years
* ongoing serious somatic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Health Anxiety Inventory (HAI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in HAI at post-treatment and follow-ups compared to baseline

SECONDARY OUTCOMES:
Illness attitude scale (IAS) | baseline, post-treatment (12 weeks), 6-month follow-up, 12-month follow-up
  Change in IAS at post-treatment and follow-ups compared to baseline
Whiteley Index (WI) | baseline, post-treatment (12 weeks) 6-month follow-up, 12 month follow-up
  Change in WI at post-treatment and follow-ups compared to baseline
Montgomery Åsberg depression rating scale-self report (MADRS-S) | baseline, post-treatment (12 weeks), 6-month follow-up, 12-month follow-up
  Change in MADRS-S at post-treatment and follow-ups compared to baseline.
Beck Anxiety Inventory (BAI) | baseline, post-treatment (12 weeks ), 6-month week follow-up, 12-month follow-up
  Change in BAI at post-treatment and follow-ups compared to baseline.
Anxiety Sensitivity Index (ASI) | baseline, post-treatment (12 weeks), 6-month follow-up, 12-month follow-up
  Change in ASI at post-treatment and follow-ups compared to baseline
Insomnia severity index (ISI) | baseline, post-treatment (12 weeks) 6-month follow-up, 12-month follow-up
  Change in ISI at post-treatment and follow-ups compared to baseline
Sheehan disability scale (SDS) | baseline, post-treatment (12) 6-month follow-up, 12-month follow-up
  Change in SDS at post-treatment and follow-ups compared to baseline
Trimbos and institute of medical technology assessment cost questionnaire (TIC-P) | baseline, post-treatment (12 weeks ), 6-month follow-up, 12-month follow-up
  Change in TIC-P at post-treatment and follow-ups compared to baseline
Euroqol-5D (EQ-5D) | baseline, post-treatment (12 weeks), 6-month follow-up, 12-month follow-up
  Change in EQ-5D)I at post-treatment and follow-ups compared to baseline
Obsessive compulsive inventory revised (OCI-R) | baseline
  Only for assessing the sample on this symptom domain at pre-treatment.
Yale-brown obsessive compulsive scale (YBOCS) | Baseline, post-treatment (variable depending on disorder), weeks 26, weeks 52
  only for assessing the sample on this domain at pre-treatment
AUDIT (alcohol use) | baseline, 12 weeks, 6 month follow-up, 12 month follow-up
  Change in AUDIT at post-treatment and follow-ups compared to baseline.

OTHER OUTCOMES:
psychological mediators | week 1, 2, 3, 4, 5, 6, 7, 8, 8, 10, 11, 12
  Assessment of whether these mediators will precede change in outcome during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, phd, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Hedman E, Andersson E, Ljotsson B, Axelsson E, Lekander M. Cost effectiveness of internet-based cognitive behaviour therapy and behavioural stress management for severe health anxiety. BMJ Open. 2016 Apr 25;6(4):e009327. doi: 10.1136/bmjopen-2015-009327. PMID 27113231
- [Derived] Hedman E, Axelsson E, Gorling A, Ritzman C, Ronnheden M, El Alaoui S, Andersson E, Lekander M, Ljotsson B. Internet-delivered exposure-based cognitive-behavioural therapy and behavioural stress management for severe health anxiety: randomised controlled trial. Br J Psychiatry. 2014 Oct;205(4):307-14. doi: 10.1192/bjp.bp.113.140913. Epub 2014 Aug 7. PMID 25104835